CLINICAL TRIAL: NCT00511511
Title: Angiogenesis Inhibitors and Hypertension: Clinical Aspects
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Other Study IDs: MEC-2007-155; EudraCT-number: 2007-002038-13
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2009-07

CONDITIONS: Hypertension
Keywords: hypertension; angiogenesis inhibitors; tyrosine kinase inhibitor; Sunitinib
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to find simple clinical and laboratory parameters to predict the development of hypertension and to elucidate the mechanism of hypertension during treatment with the tyrosine kinase inhibitor Sunitinib.

DETAILED DESCRIPTION:
Inhibition of angiogenesis with antibodies against vascular endothelial growth factor (VEGF) and VEGF receptor antagonists has become an established treatment for cancer. An unanticipated side effect of angiogenesis inhibitors is the development of hypertension. The pathogenesis of this hypertension is unknown. Not all patients will develop hypertension. However, it is not known which patient will and which patient will not develop hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, with either renal cell carcinoma or gastro intestinal stromal tumors (GIST) intended to be treated solely with Sunitinib (single-agent treatment) and who are considered fit enough by their treating physician to receive Sunitinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women, with either renal cell carcinoma or gastro intestinal stromal tumors (GIST) intended to be treated solely with Sunitinib (single-agent treatment) and who are considered fit enough by their treating physician to receive Sunitinib
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2007-08; Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. H. van den Meiracker, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

REFERENCES:
- [Background] Zakarija A, Soff G. Update on angiogenesis inhibitors. Curr Opin Oncol. 2005 Nov;17(6):578-83. doi: 10.1097/01.cco.0000183672.15133.ab. PMID 16224236
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Miller KD, Chap LI, Holmes FA, Cobleigh MA, Marcom PK, Fehrenbacher L, Dickler M, Overmoyer BA, Reimann JD, Sing AP, Langmuir V, Rugo HS. Randomized phase III trial of capecitabine compared with bevacizumab plus capecitabine in patients with previously treated metastatic breast cancer. J Clin Oncol. 2005 Feb 1;23(4):792-9. doi: 10.1200/JCO.2005.05.098. PMID 15681523
- [Background] Sica DA. Angiogenesis inhibitors and hypertension: an emerging issue. J Clin Oncol. 2006 Mar 20;24(9):1329-31. doi: 10.1200/JCO.2005.04.5740. Epub 2006 Jan 30. No abstract available. PMID 16446321
- [Background] Veronese ML, Mosenkis A, Flaherty KT, Gallagher M, Stevenson JP, Townsend RR, O'Dwyer PJ. Mechanisms of hypertension associated with BAY 43-9006. J Clin Oncol. 2006 Mar 20;24(9):1363-9. doi: 10.1200/JCO.2005.02.0503. Epub 2006 Jan 30. PMID 16446323
- [Background] Deanfield JE, Halcox JP, Rabelink TJ. Endothelial function and dysfunction: testing and clinical relevance. Circulation. 2007 Mar 13;115(10):1285-95. doi: 10.1161/CIRCULATIONAHA.106.652859. No abstract available. PMID 17353456
- [Background] Kuenen BC, Levi M, Meijers JC, Kakkar AK, van Hinsbergh VW, Kostense PJ, Pinedo HM, Hoekman K. Analysis of coagulation cascade and endothelial cell activation during inhibition of vascular endothelial growth factor/vascular endothelial growth factor receptor pathway in cancer patients. Arterioscler Thromb Vasc Biol. 2002 Sep 1;22(9):1500-5. doi: 10.1161/01.atv.0000030186.66672.36. PMID 12231573
- [Background] Bosnjak JJ, Terata K, Miura H, Sato A, Nicolosi AC, McDonald M, Manthei SA, Saito T, Hatoum OA, Gutterman DD. Mechanism of thrombin-induced vasodilation in human coronary arterioles. Am J Physiol Heart Circ Physiol. 2003 Apr;284(4):H1080-6. doi: 10.1152/ajpheart.00465.2002. Epub 2002 Dec 19. PMID 12595282
- [Background] Touyz RM. Regulation of endothelial nitric oxide synthase by thrombin. Hypertension. 2007 Mar;49(3):429-31. doi: 10.1161/01.HYP.0000255955.75119.1a. Epub 2007 Jan 8. No abstract available. PMID 17210837
- [Background] Ferrara N, Gerber HP, LeCouter J. The biology of VEGF and its receptors. Nat Med. 2003 Jun;9(6):669-76. doi: 10.1038/nm0603-669. PMID 12778165
- [Background] Henry TD, Annex BH, McKendall GR, Azrin MA, Lopez JJ, Giordano FJ, Shah PK, Willerson JT, Benza RL, Berman DS, Gibson CM, Bajamonde A, Rundle AC, Fine J, McCluskey ER; VIVA Investigators. The VIVA trial: Vascular endothelial growth factor in Ischemia for Vascular Angiogenesis. Circulation. 2003 Mar 18;107(10):1359-65. doi: 10.1161/01.cir.0000061911.47710.8a. PMID 12642354
- [Background] Hood JD, Meininger CJ, Ziche M, Granger HJ. VEGF upregulates ecNOS message, protein, and NO production in human endothelial cells. Am J Physiol. 1998 Mar;274(3):H1054-8. doi: 10.1152/ajpheart.1998.274.3.H1054. PMID 9530221
- [Background] Li B, Ogasawara AK, Yang R, Wei W, He GW, Zioncheck TF, Bunting S, de Vos AM, Jin H. KDR (VEGF receptor 2) is the major mediator for the hypotensive effect of VEGF. Hypertension. 2002 Jun;39(6):1095-100. doi: 10.1161/01.hyp.0000018588.56950.7a. PMID 12052848
- [Background] Broere A, Van Den Meiracker AH, Boomsma F, Derkx FH, Veld AJ, Schalekamp MA. Human renal and systemic hemodynamic, natriuretic, and neurohumoral responses to different doses of L-NAME. Am J Physiol. 1998 Dec;275(6):F870-7. doi: 10.1152/ajprenal.1998.275.6.F870. PMID 9843903
- [Background] van der Linde NA, Boomsma F, van den Meiracker AH. Role of nitric oxide in modulating systemic pressor responses to different vasoconstrictors in man. J Hypertens. 2005 May;23(5):1009-15. doi: 10.1097/01.hjh.0000166842.65097.b1. PMID 15834287
- [Derived] Kappers MH, van Esch JH, Sluiter W, Sleijfer S, Danser AH, van den Meiracker AH. Hypertension induced by the tyrosine kinase inhibitor sunitinib is associated with increased circulating endothelin-1 levels. Hypertension. 2010 Oct;56(4):675-81. doi: 10.1161/HYPERTENSIONAHA.109.149690. Epub 2010 Aug 23. PMID 20733093